CLINICAL TRIAL: NCT00211796
Title: Divalproex Sodium ER in Adult Autism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Eric Hollander, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO#04-1106
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Autism
Keywords: autism; divalproex sodium ER; aggression; irritability
MeSH Terms: conditions — Autistic Disorder; Aggression

INTERVENTIONS:
Drug: Divalproex Sodium ER

SUMMARY:
12-week open label treatment trial of divalproex sodium extended release (Depakote ER) in 10 patients with a diagnosis of autism. Our objective is to determine how well these patients can tolerate the prescribed doses and what added benefits can be attributed to divalproex sodium ER.

DETAILED DESCRIPTION:
Based on positive research with divalproex in children/adolescents with autism, we would like to extend this research to autistic adults with high levels of aggression, irritability, affective instability, or agitation. We aim to have 10 adult autistic patients enrolled in our study of the treatment of aggression/irritability with divalproex sodium ER. This will be an open treatment for adult patients to determine if the tolerability of divalproex sodium is better with the extended release. We propose this open label design because previous double-blinded studies of divalproex sodium were only done in children, not adults. These results will serve as pilot data for a future blinded study for autistic adults with the extended release formulation. This naturalistic design will allow for prior stable (3 months) use of concomitant medications. Our objective is to determine how well these patients can tolerate the prescribed doses and what added benefits can be attributed to divalproex sodium ER.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV, ADI, or ADOS criteria for autism spectrum disorder.
2. Age 18-65.
3. Be seen as outpatients
4. Demonstrate capacity to provide authorized informed consent or provide consent for participation by an approved surrogate on the autistic individual's behalf
5. Sexually active females of childbearing potential must use an acceptable method of birth control and have a negative serum pregnancy test prior to entry into the study.
6. Score at least 4 (moderately ill) on the Clinical Global Impression-Severity Scale for Autistic Disorder (CGI-AD).
7. Subject meets the following criteria at pre-study diagnostic assessment and baseline assessment: OAS-M 6 (raw scores).
8. Subjects on a stable dose of their current psychotropic medication for at least 3 months before entering the study, with the understanding that they must remain on a stable dose throughout the trial. If a subject chooses to taper off their current medications, they will be closely monitored by the study psychiatrist and must be medication free for 2 weeks prior to beginning the study. Additionally, if a subject is currently taking a medication with a known drug interaction with Divalproex Sodium, he/she will be tapered off of that medication under the supervision of the study psychiatrist before undergoing treatment.

Exclusion Criteria:

1. Subjects who are pregnant or nursing mothers. Sexually active women of childbearing potential who are not using adequate birth control measures.
2. Subjects with active or unstable epilepsy.
3. Subjects with any of the following past or present mental disorders: schizophrenia, schizoaffective disorder, bipolar disorder, or organic mental disorders.
4. Subjects who are a serious suicidal risk.
5. Subjects with clinically significant or unstable medical illness that would contraindicate participation in the study, including hematopoietic or cardiovascular disease, pancreatitis, liver toxicity, and polycystic ovary syndrome.
6. Subjects reporting history of encephalitis, phenylketonuria, tuberous schelrosis, fragile X syndrome, anoxia during birth, pica, neurofibromatosis, hypomelanosis of Ito, hypothyroidism, Duchenne muscular dystrophy, and maternal rubella.
7. Patients with history of the following:

   * gastrointestinal, liver, or kidney, or other known conditions which will presently interfere presently with the absorption, distribution, metabolism, or excretion of drugs.
   * cerebrovascular disease or brain trauma
   * clinically significant unstable endocrine disorder, such as hypo- or hyperthyroidism
   * recent history or presence of any form of malignancy
   * Subjects with an unstable history of seizures cannot participate in the study. However, subjects who have been seizure-free for at least 6 months on a stable dose of anticonvulsant medication other than divalproex sodium or related formulations (e.g., depakene) may participate, along with non-medicated subjects with a history of seizures who have been seizure-free for at least 6 months. Subjects with abnormal EEG but no clinical seizures are also eligible.
8. Treatment within the previous 30 days with any drug known to a well-defined potential for toxicity to a major organ
9. Subjects with clinically significant abnormalities in laboratory tests or physical exam.
10. Subjects with a history of hypersensitivity or severe side effects associated with the use of divalproex sodium, or other an ineffective prior therapeutic trial of divalproex sodium (serum levels within range of 50-100 ug/ml for 6 weeks).
11. Subjects who are currently taking a medication with a known drug interaction with Divalproex Sodium (betamipron, chaparral, cholestyramine, clarithromycin, comfrey, ethosuximide, evening primrose, felbamate, fosphenytoin, germander, ginkgo, jin bu huan, kava, mefloquine, panipenem, pennyroyal, primidone, rifampin, rifapentine, and zidovudine) and refuse to taper off of that medication.
12. Subjects who are already being treated with Divalproex Sodium.
13. Subjects with any organic or systemic disease or patients who require a therapeutic intervention, not otherwise specified, which would confound the evaluation of the safety of the study medication.
14. Subjects who reside in a remote geographical area who do not have regular access to transportation to the clinical facility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
the Clinical Global Improvement and Severity scales (CGI-I and CGI-S)
Overt Aggression Scale-Modified (OAS M)
Affective Lability Scale (ALS).

SECONDARY OUTCOMES:
Global Assessment of Functioning Scale (GAF)
Aggression Questionnaire (AQ)
the Hamilton Depression (Ham-D) Scale
Yale Brown Obsessive Compulsion Scale (YBOCS)
Compulsion sub-scale
Aberrant Behavior Checklist (ABC)
Barratt Impulsiveness Scale
Version11 (BIS-11).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States